CLINICAL TRIAL: NCT02706353
Title: Phase I/II Dose Escalation and Cohort Expansion of Safety and Tolerability Study of Intratumoral CD40 Agonistic Monoclonal Antibody APX005M in Combination With Systemic Pembrolizumab in Patients With Metastatic Melanoma
Brief Title: APX005M in Combination With Systemic Pembrolizumab in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: <75% participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Apexigen America, Inc. (Industry); Pyxis Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0654; NCI-2016-00675 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic Melanoma; Intratumoral APX005M; Pembrolizumab; Keytruda; MK-3475; SCH-900475
MeSH Terms: conditions — Melanoma | interventions — sotigalimab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APX005M + Pembrolizumab (Experimental): Dose Escalation Phase:
  Starting dose level of APX005M is 0.1 mg injected directly into 1-3 tumors every 3 weeks (Weeks 0, 3, 6, and 9) for up to 4 doses. Tumor site chosen based on volume to be injected.
  All participants receive Pembrolizumab at 2 mg/kg by vein 1 time every 3 weeks (Weeks 0, 3, 6, 9, and 12). First dose of Pembrolizumab given 1-2 days before or after first dose of APX005M.
  Dose Expansion Phase:
  Starting dose level of APX005M is maximum tolerated dose from Dose Escalation Phase.
  Participants receive same dosage of Pembrolizumab as in Dose Escalation Phase.
  Interventions: Drug: APX005M; Drug: Pembrolizumab

INTERVENTIONS:
Drug: APX005M — Dose Escalation Phase Starting Dose Level of APX005M: 0.1 mg injected directly into 1-3 tumors every 3 weeks (Weeks 0, 3, 6, and 9) for up to 4 doses.
  Dose Expansion Phase Starting Dose Level of APX005M: Maximum tolerated dose from Dose Escalation Phase.
Drug: Pembrolizumab — Dose Escalation and Expansion Phase Dose of Pembrolizumab: 2 mg/kg by vein 1 time every 3 weeks (Weeks 0, 3, 6, 9, and 12). First dose of Pembrolizumab given 1-2 days before or after first dose of APX005M.
  Other Names: Keytruda; MK-3475; SCH-900475

SUMMARY:
You are being asked to take part in this study because you have metastatic (cancer that has spread) melanoma.

The goal of Part 1 of this clinical research study is to find the highest tolerable dose of APX005M that can be given with pembrolizumab that can be given to patients with metastatic melanoma.

The goal of Part 2 of this study is to learn if the combination can help to control metastatic melanoma.

The safety of this drug combination will also be studied.

This is an investigational study. APX005M is not FDA approved or commercially available. It is currently being used for research purposes only. Pembrolizumab is FDA approved and commercially available for the treatment of metastatic melanoma. The combination of these drugs to treat metastatic melanoma is investigational.

The study doctor can explain how the study drug is designed to work.

Up to 41 participants will be treated in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of 3 participants will be enrolled in Part 1, and up to 20 participants will be enrolled in Part 2.

If you are enrolled in Part 1, the dose of APX005M you receive will depend on when you join this study. The first group of participants will receive the lowest dose level of APX005M. Each new group will receive a higher dose of APX005M than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of APX005M is found.

If you are enrolled in Part 2, you will receive APX005M at the highest dose that was tolerated in Phase 1

All participants will receive the same dose level of pembrolizumab.

Study Drug Administration:

APX005M will be injected directly into 1 tumor every 3 weeks (Weeks 0, 3, 6, and 9) for up to 4 doses.

The injections may be done with or without the help of a ultrasound, CT, and MRI.

If the doctor thinks it is needed, you may need to stay in the hospital overnight or be monitored by a caregiver for 24 hours after you receive APX005M.

You will receive pembrolizumab by vein 1 time every 3 weeks (Weeks 0, 3, 6, 9, and 12). The first dose of pembrolizumab will be given 1-2 days before or after your first dose of APX005M.

You will be given a diary to write down any injection site reactions you may have.

Study Visits:

Within 1 week before your first APX005M injection:

* You will have a physical exam.
* You will have a punch biopsy or image-guided biopsy of a tumor to check the status of the disease. To collect a biopsy, the area of skin is numbed with anesthetic and a small cut is made to remove all or part of the affected tissue. To collect a punch biopsy, the area of skin is numbed with anesthetic and a small cut is made to remove all or part of the affected tissue. To perform an image-guided biopsy, a needle is inserted into the affected area using imaging such as CT or ultrasound to collect cells or tissue from an organ, lymph node, or suspected tumor mass. The doctor will use the imaging to guide the needle into the area.
* Blood (about 4½ tablespoons) will be drawn to test your immune system. If you can become pregnant, blood (about 1 teaspoon) may be drawn for a pregnancy test or urine may be collected to test for pregnancy.
* The tumors may be measured and photographed.

On Day 1 of Cycle 1:

* You will have a physical exam.
* Blood (about 5½ tablespoons) will be drawn for routine tests and test your immune system.
* The tumor may be measured and photographed.

On Day 2 of Cycle 1:

* Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have a biopsy of one of the injected tumor sites within about 24 hours after the 1st injection to check the status of the disease.

On Day 3 of Cycle 1:

* Your vital signs will be measured.
* Blood (about 5 tablespoons) will be drawn for routine tests and to test your immune system.

On Days 8 and 15 of Cycle 1:

* Your vital signs will be measured.
* Blood (about 1½ teaspoons) will be drawn for routine tests.
* Blood (about 4½ tablespoons) may be drawn to test your immune system (Day 8 only).

On Day 1 of Cycle 2:

* You will have a physical exam.
* Blood (about 5½ tablespoons) will be drawn for routine tests and to test your immune system.

On Days 8 and 15 of Cycle 2:

* Your vital signs will be measured.
* Blood (about 1½ teaspoons) will be drawn for routine tests.
* Blood (about 4½ tablespoons) may be drawn to test your immune system (Day 8 only).

On Day 1 of Cycle 3 (± 3 days):

* Your vital signs will be measured.
* You will have a physical exam.
* You will have a biopsy of one of the injected tumors and one of the tumors for which you did not have an injection to check the status of the disease.
* The tumors may be measured and photographed.
* You will have CT, MRI/CT, and/or an ultrasound to check the status of the disease.
* Blood (about 2½ teaspoons) will be drawn for routine tests. If you can become pregnant, a pregnancy test may be performed. Urine may be collected for the pregnancy test.
* Blood (about 4½ tablespoons) will be drawn to test your immune system.

On Day 1 of Cycle 4:

* Your vital signs will be measured
* You will have a physical exam.
* Blood (about 2½ teaspoons) will be drawn for routine tests
* Blood (about 4½ tablespoons) will be drawn to test your immune system.

On Day 1 of Cycles 5-8:

* Your vital signs will be measured.
* You will have a physical exam.
* Blood (about 1½ teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 5 and 8 ONLY (± 3 days):

* Blood (about 1½ teaspoons) will be drawn for routine tests.
* Blood (about 4½ tablespoons) will be drawn to test your immune system.
* You may have a biopsy of one of the injected tumors and one of the tumors for which you did not have an injection to check the status of the disease (Cycle 5 only).
* The tumors may be measured and photographed.
* You will have CT, MRI/CT, and/or an ultrasound to check the status of the disease.

Cycles beyond Cycle 8:

°You will have CT, MRI/CT, and/or an ultrasound to check the status of the disease (every 3 months for up to 2 years).

Length of Treatment:

You will be on study for up to 2 years. You will be taken off study if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

If your doctor thinks it is in your benefit, you may continue to receive pembrolizumab as standard of care after you are off this study. Your doctor will describe this in more detail.

Off-Study Visit:

If you have to go off study early because the disease got worse or you had intolerable side effects:

* Your vital signs will be measured.
* You will have a physical exam.
* Blood (about 1½ teaspoons) will be drawn for routine tests.
* Blood (about 4½ tablespoons) will be drawn to test your immune system.

Follow-Up:

Within 2 weeks after your last study drug dose and every 8-12 weeks after that, you may have scans to check the status of the disease. Your doctor will decide what type of scans you will have.

If you choose to seek care at another hospital, the study staff will call you every 3 months for up to 2 years after your last study drug dose. You will be asked how you are doing. The calls should last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Histologically or cytologically confirmed malignant melanoma from skin, or mucosal melanoma (i.e. ocular melanoma subjects are not eligible)
3. Measurable, unresectable stage III (in transit lesions) or stage IVA, IVB, IVC disease
4. At least two injectable lesions (amenable for direct injection or through the use of image guidance such ultrasound [US], CT or MRI) defined as any injectable cutaneous, subcutaneous, nodal, or visceral melanoma lesion ≥ 10 mm in longest diameter
5. Age ≥ 18 years
6. ECOG performance status 0 or 1
7. Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
8. Platelet count greater than or equal to 100,000/mm^3
9. WBC >3000/mm^3
10. ANC > 1500/mm^3
11. Hemoglobin >9 g/dL
12. Serum ALT and AST <3 the upper limit of normal (ULN); <5 ULN if there is liver involvement secondary to the tumor
13. Serum creatinine < 2.0 mg/dl
14. Seronegative for HIV antibody
15. Patients with a negative pregnancy test (urine or serum) must be documented within 14 days of screening for women of childbearing potential (WOCBP). A WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e. who has not had menses at any time in the preceding 12 consecutive months). Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the patient agrees to continue to use a barrier method of contraception throughout the study and for 4 months after the last dose of APX005M or Pembrolizumab such as: condom, diaphragm, hormonal, IUD, or sponge plus spermicide. Abstinence is an acceptable form of birth control.

Exclusion Criteria:

1. Patients who have previously received pembrolizumab or PD-/L1 blockade therapy. Adjuvant IFN-a, is allowed if last dose was received at least 6 months of starting study treatment.
2. Active autoimmune disease requiring disease-modifying therapy.
3. Concurrent systemic steroid therapy higher than physiologic dose (>7.5 mg/day of prednisone or equivalent).
4. Any form of active primary or secondary immunodeficiency.
5. History of hematologic malignancy.
6. Active coagulopathy.
7. History of New York Heart Association class 3-4 congestive heart failure or history myocardial infarction within 6 months of starting study treatment.
8. History of arterial thrombosis within 3 months of starting study treatment.
9. Patients with known symptomatic brain metastases requiring systematic corticosteroids. Patients with previous diagnosed brain metastases are eligible if they have completed their treatment and have recovered from acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for their metastases for at least 2 weeks and are neurologically stable. Mild neurological deficits are allowed, if they do not interfere with the ability to judge the safety profile of APX005M.
10. Prior malignancy except the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, thyroid cancer (except anaplastic) or any cancer from which the patient has been disease-free for 2 years.
11. Subjects who have received prior immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1), anti-CD40.
12. Subjects that have received experimental vaccines or other immune therapies should be discussed with the Principal Investigator to confirm eligibility.
13. Active known clinically serious infections (> Grade 2 NCI-CTCAE version 4.03).
14. Prior systemic therapy, radiation therapy, or surgery within the 28 days of starting study treatment. Palliative radiotherapy to a limited field or palliative cryoablation is allowed after consultation with the Principal Investigator, at any time during the study participation including screening.
15. Women of child-bearing potential (WOCBP), women who are pregnant, or women who are nursing.
16. Known or underlying medical condition that, in the opinion of the investigator or sponsor, could make the administration of study drug hazardous to the subjects, or could adversely affect the ability of the subject to comply with or tolerate study procedures and/or study therapy, or confound the ability to interpret the tolerability of combined administration of APX005M and Pembrolizumab in treated subjects.
17. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
18. Has received a TB skin test within 14 days before the first dose of study drug.
19. Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adi Diab, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dose Escalation and Cohort Expansion of Safety and Tolerability of Intratumoral CD40 Agonistic Monoclonal Antibody APX005M in Combination with Systemic Pembrolizumab.
Pre-assignment Details: 40 subjects consented; 6 pts not eligible; 32 subjects treated & 2 subjects in the Expansion Phase withdrew consent prior to screening assessments
Groups:
- Phase 1: Dose Escalation (0.1 mg): IT APX005M DL 1-DL 5 0.1 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks
  Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 1: Dose Escalation (0.5 mg): IT APX005M DL 1-DL 5 0.5 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks
  Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 1: Dose Escalation (1 mg): IT APX005M DL 1-DL 5 1 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks
  Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 1: Dose Escalation (3 mg): IT APX005M DL 1-DL 5 3 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks
  Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 1: Dose Escalation (10 mg): IT APX005M DL 1-DL 5 10 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks
  Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 2: Dose Expansion: IT APX005M 10 mg q3 wks & Pembrolizumab IV 200 mg (flat dose) q3 wks
Period: Dose Level 1
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Started | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Started | 0 | 1 | 0 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Started | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 2 | 0 | 0 | 0
Period: Dose Level 4
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Started | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Toxicity | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Period: Dose Level 5
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Started | 0 | 0 | 0 | 0 | 6 | 20
Completed | 0 | 0 | 0 | 0 | 1 | 10
Not Completed | 0 | 0 | 0 | 0 | 5 | 10
Not completed — Toxicity | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Dose Escalation: IT APX005M DL 1-DL 5 0.1 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks
  Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Escalation | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 20 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 1 | 2 | 13 | 18
  >=65 years | 1 | 0 | 2 | 2 | 4 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 4 | 7
  Male | 1 | 1 | 2 | 3 | 4 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 0 | 1 | 3 | 2 | 6 | 18 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 0 | 1 | 3 | 3 | 5 | 19 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 3 | 3 | 6 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: To assess safety and tolerability of intratumoral APX005M given with systemic pembrolizumab and identify of the maximum tolerated dose/recommended phase 2 dose (MTD/PR2D) of the combination therapy in patients with metastatic melanoma.
Time Frame: Baseline to 2 years
Measure: Number; unit: mg
Arm/Group | Phase 1: Dose Escalation | Phase 2: Dose Expansion
Number analyzed (Participants) | 14 | 18
mg | 10 | 10

2. Primary Outcome: Overall Response Rate (ORR)
Description: To assess best overall response after ibtratumoral injection of APX005M in combination with systemic pembrolizumab
Time Frame: Baseline to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 18
percentage of participants | 0 | 0 | 33.3 | 66.7 | 50 | 50

3. Secondary Outcome: Evaluation of Intratumoral CD8⁺ T Cells
Description: To comprehensively assess CD8⁺ T cell responses in injected tumors, we employed multiplex immunofluorescence (mIF).
Time Frame: Baseline to week 6
Population: Although 32 patients were enrolled in the study, only 26 were included in the biomarker analyses. The remaining 6 were excluded due to issues such as insufficient or poor-quality tumor tissue and/or the absence of paired tumor samples necessary for direct comparisons.
Measure: Mean (Standard Deviation); unit: density cells/mm^2
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 6 | 13
density cells/mm^2 | 12.04 | 1409.18 | -24.62 (42.21) | 17.60 (68.98) | 415.92 (695.56) | 388.1 (435.1)

4. Secondary Outcome: Overall Safety and Tolerability
Description: To assess the overall safety and tolerability of IT APX005M given with systemic pembrolizumab in patients with metastatic melanoma.
Time Frame: Baseline to 2 years
Measure: Number; unit: grade 3/grade 4 events
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 18
grade 3/grade 4 events | 0 | 1 | 1 | 12 | 5 | 28

5. Secondary Outcome: Anti-tumor Immune Responses and Clinical Efficacy
Description: To evaluate anti-tumor immune responses and clinical efficacy of intratumoral injection of IT APX005M with systemic Pembrolizumab
Time Frame: Baseline to 2 years
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1: Dose Escalation (0.01 mg): T APX005M DL 1-DL 5 0.1 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 1: Dose Escalation (1 mg): T APX005M DL 1-DL 5 0.5 mg q3 wks & Pembrolizumab 2 mg/kg (mas 200 mg) q3 wks Dose level 1 = 0.1 mg Dose level 2 = 0.5 mg Dose level 3 = 1 mg Dose level 4 = 3 mg Dose level 5 = 10 mg
- Phase 2: intratumoral APX005M at the RP2D with pembrolizumab
Arm/Group | Phase 1: Dose Escalation (0.01 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 18
percentage of participants | 0.00 [0.00 to 98.80] | 0.00 [0.00 to 98.80] | 33.3 [0.40 to 93.40] | 66.70 [6.60 to 99.60] | 50.00 [9.20 to 90.80] | 50.00 [23.40 to 76.60]

ADVERSE EVENTS:
Time Frame: Baseline to 2 years
Arm/Group | Phase 1: Dose Escalation (0.1 mg) | Phase 1: Dose Escalation (0.5 mg) | Phase 1: Dose Escalation (1 mg) | Phase 1: Dose Escalation (3 mg) | Phase 1: Dose Escalation (10 mg) | Phase 2: Dose Expansion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 1/3 | 1/6 | 6/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 1/3 | 1/6 | 9/20
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 6/6 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation (0.1 mg) (N=1) | Phase 1: Dose Escalation (0.5 mg) (N=1) | Phase 1: Dose Escalation (1 mg) (N=3) | Phase 1: Dose Escalation (3 mg) (N=3) | Phase 1: Dose Escalation (10 mg) (N=6) | Phase 2: Dose Expansion (N=20)
Intra-abdominal hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal hiatial hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Saddle PE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infaraction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromeoemeolic Event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation (0.1 mg) (N=1) | Phase 1: Dose Escalation (0.5 mg) (N=1) | Phase 1: Dose Escalation (1 mg) (N=3) | Phase 1: Dose Escalation (3 mg) (N=3) | Phase 1: Dose Escalation (10 mg) (N=6) | Phase 2: Dose Expansion (N=20)
Fatigue (General disorders) | 0 (0) | 1 | 2 (2) | 2 (6) | 2 (4) | 14 (25)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (7) | 6 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (18)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sigmoid diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Edema- injection site (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hip pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 7 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 2 (4) | 3 (24) | 5 (18) | 14 (32)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 3 (7) | 7 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (2) | 6 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (12) | 2 (3) | 11 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 8 (15)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Infection Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis prophylaxis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection Oral Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (33)
Infusion related action (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 5 (15) | 13 (40)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Left knee swollen (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and Connective Tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 7 (10)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 3 (4)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain inextremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bilateral peripheral neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 2 (2) | 1 (3) | 3 (15) | 7 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (19) | 4 (5)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Redness in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (5)
Watery eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Right shoulder injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Prothromibn Time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALK decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (14) | 3 (8)
Injection site - redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Warmth-Injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (19) | 1 (2)
Skin injection site pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Skin-benign nevi (trunk) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin-actinic keratosis (left dorsal hand) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin-lichenoid dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin redness-lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin-lichenoid reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin-vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Non-inflamed seborrheic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lentigines and cherry angioma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pigmented macules (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma in situ (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Redness tumor injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Skin warmth (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin rash on chest and arm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczematous Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflamed seborrheic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Heat exhaustion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 3 (16)
Left axilla pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Left axilla -differential diagnosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laparoscopy hernia repair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain-surgical site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin-Rash, contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chondrodermatitis nodularis helicis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blistering at tape site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin redness with blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nummular dermatitis - pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alamine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 4 (9) | 12 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 3 (7) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (15) | 4 (7) | 14 (29)
Chelitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Alakaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (3) | 6 (7)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 3 (4) | 0 (0)
Brusing (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (9) | 4 (5)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 5 (10) | 9 (19)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 3 (8) | 8 (12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 3 (4)
Skin-lichenoid (central chest) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (3) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal TSH (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Alopcia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asparatate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (17)
Blood and lymphatic systems disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Elevated TSH (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Congenital retainal pigment epithelial hypertrophy rt. eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right lung pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthrodism- elevated TSH (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritic rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Plantar facitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT02706353/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT02706353/ICF_001.pdf